CLINICAL TRIAL: NCT06828770
Title: Post-Approval Study of the Renata Minima Stent in the Treatment of Vascular Stenoses in Neonates, Infants, and Small Children
Brief Title: Minima Stent System Post- Approval Study (PAS)
Status: Recruiting | Type: Observational
Sponsor: Renata Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: PTC-0038
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Artery Stenosis; Aortic Coarctation
Keywords: Vascular Stenosis; Minima; Minima Stent; Minima Stent System; Renata Medical; Renata; infant stent
MeSH Terms: conditions — Stenosis, Pulmonary Artery; Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Minima PAS Patients: Those treated with the Renata Minima Stent System
  Interventions: Device: Minima Stent System

INTERVENTIONS:
Device: Minima Stent System — Minima Stent System is indicated for use in the treatment of native or acquired pulmonary artery stenoses or coarctation of the aorta in neonates, infants, and children at least 1.5kg in weight.

SUMMARY:
This Post-Approval Study is a single arm, prospective, multi-center, open-label study of patients treated with the Renata Minima Stent System in the United States. The objective of the study is to continue the assessment of device performance and capture outcome data on use of the device in real-world use.

DETAILED DESCRIPTION:
A minimum of 100 subjects will be enrolled. Follow-up will occur immediately after the initial implant procedure, at subsequent re-dilation procedures, annually, and at any additional standard of care follow-up visits (determined by the implanting physician) through 5 years post-implant. Data collected at each follow-up will be used in analysis. This study will monitor key data points related to the device and procedure.

ELIGIBILITY:
Inclusion Criteria:

* The subject's legally authorized representative has been informed of the nature of the device treatment, agrees to its provisions, and has provided written informed consent
* Indicated for treatment with the Minima Stent System per the IFU.

Exclusion Criteria:

* Active bloodstream infection requiring antibiotic therapy within 3 days prior to stent implantation
* History of or active endocarditis (active treatment with antibiotics) within 180 days prior to stent implantation
* Aortic or pulmonary artery aneurysm in the location targeted for treatment
* Body weight < 1.5 kg
* Anatomic location of lesion judged by the investigator to not lend to the safe placement of a stent
* Target vessels larger or smaller than the Minima System balloon size ranges
* Known genetic syndrome known to be associated with vasculopathies such as but not limited to Williams syndrome, Loeys-Dietz syndrome, etc
* Clinical scenario requiring that more than one vessel needs stent implantation at the time of the trial procedure.
* Currently participating in an investigational drug study or another device study
* Major or progressive non-cardiac disease resulting in a life expectancy of less than six months
* Known hypersensitivity to aspirin or heparin and cannot be treated with other antiplatelet and/or antithrombotic medications
* Known hypersensitivity to cobalt-chromium or contrast media that cannot be adequately premedicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with the Renata Minima Stent System in the United States
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Acute Device Success | End of Procedure (Following Implantation of the Stent)
  Rate of Acute device success as defined by:
  * Stenosis relief, defined by stent outer diameter ≥ 75% of the normal surrounding vessel immediately after deployment.
  * Freedom from open surgical intervention required to treat Minima Stent dysfunction at implantation
Rate of Participants with Freedom from procedure- or device-related SAEs | Immediately after Postoperative
  Rate of Participants with Freedom from procedure- or device-related SAEs resulting in an event listed below:
  * Death
  * Cardiac arrest and/or emergency ECMO cannulation
  * Stroke
  * Limb loss
  * Vessel dissection of target lesion
  * Device thrombosis/occlusion
  * Cardiac perforation requiring percutaneous or open surgical intervention
  * Persistent cardiac arrhythmia requiring a pacemaker

SECONDARY OUTCOMES:
Rate of Successful Stent Re-Dilation and Peak-to-Peak Pressure gradient | During and end of procedure
  * Peak-to-peak pressure gradient (ventricle to arterial or arterial to arterial) < 20 mmHg after stent placement, in treatment of Aortic Coarctation, when applicable.
  * Successful stent re-dilation (when indicated) at recatheterization, defined as angiographic improvement of stenosis to >50% of the normal surrounding vessel.
  * Maintenance of stented vessel diameter ≥ 50% of post implant diameter at the time of re-dilation (pre re-dilation).
Rate of Participants with Freedom from Stent Migration/Embolization, procedure- or device- related SAEs, and non-elective stent explant | During and at end of procedure
  * Freedom from intraprocedural stent movement to non-intended location during the procedure.
  * Freedom from postprocedural stent embolization or migration
  * Freedom from stent fracture that led to reintervention
  * Freedom from non-elective Minima Stent explant
  * Freedom from procedure- or device-related SAE during re-dilation that results in the following:
    * Death
    * Cardiac arrest and/or emergency ECMO cannulation
    * Stroke
    * Limb loss
    * Vessel dissection of target lesion
    * Device thrombosis/occlusion
    * Cardiac perforation requiring percutaneous or open surgical intervention
    * Persistent cardiac arrhythmia requiring a pacemaker

CONTACTS AND LOCATIONS:
Overall Officials: Arash Salavitabar, MD, Principal Investigator — Nationwide Children's Hospital
Locations (15):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, Saint Louis, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Dell Children's Medical Center, The University of Texas at Austin, Austin, Texas
  - Columbia Hospital at Medical City Dallas Hospital, Dallas, Texas
  - UVA Health Children's Hospital, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No